CLINICAL TRIAL: NCT06818799
Title: Evaluation of Thulium Laser Endoscopic En-bloc Resection Versus Conventional Trans-urethral En-bloc Resection of Primary Non-muscle Invasive Bladder Cancer
Brief Title: Thulium Laser En-bloc Resection of Primary Non-muscle Invasive Bladder Cancer
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Helwan University (Other)
Collaborators: Ain Shams University (Other); Maadi Military Hospital (Other Government)
Responsible Party: Principal Investigator, Samuel Fayek Tawfeles Ebskharoun, Principal investigator, Helwan University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 82-2023
Record Dates: First submitted 2025-02-05; First posted 2025-02-10 (Actual); Last update posted 2025-02-12 (Actual); Status verified 2025-02

CONDITIONS: Bladder Transitional Cell Carcinoma
Keywords: Thulium laser resection of bladder mass; Trans-urethral resection of bladder mass; Non muscle-invasive bladder cancer
MeSH Terms: conditions — Non-Muscle Invasive Bladder Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Thulium laser "TmLRBT" (Experimental): Participants recieved thulium laser en-bloc resection of bladder mass
  Interventions: Procedure: Thulium laser en-bloc resection of bladder mass
- Trans-Urethral resection "TURBT" (Active Comparator): Participants recieved trans-urethral en-bloc resection of bladder mass
  Interventions: Procedure: Trans-urethral en-bloc resection of bladder mass

INTERVENTIONS:
Procedure: Thulium laser en-bloc resection of bladder mass — En-bloc laser technique
  Arms: Thulium laser "TmLRBT"
Procedure: Trans-urethral en-bloc resection of bladder mass — En-bloc technique
  Arms: Trans-Urethral resection "TURBT"

SUMMARY:
The goal of this clinical trial is to know if thulium laser works to treat non-muscle invasive bladder cancer "NMIBC" efficiently in comparison to classical trans-urethral resection "TURBT". It will also learn about the safety of this technique. The main questions it aims to answer are:

Does thulium laser lower the incidence of recurrence to participants with non- muscle invasive bladder cancer? What complications do participants have when using this technique? Investigators will compare thulium laser en-bloc resection to a classical trans-urethral en-bloc resection of bladder tumor

Participants will:

Do thulium laser en-bloc resection or trans-urethral en-bloc resection And will be classified to risk group according to European association of urology guidelines and followed up accordingly.

DETAILED DESCRIPTION:
The conventional transurethral resection of bladder tumor (TURBT) is the most common strategy for NMIBC and it is recommended by the guidelines. However, the TURBT has a complication rate of ~4-6%, of which urinary tract infections and significant haematuria are most common.

In some cases, major complications including obturator nerve reflex (ONR) and bladder perforation could occur. To overcome these drawbacks, lasers including holmium YAG and thulium YAG were introduced. Several studies have suggested the superior safety of Thulium laser resection of bladder tumors (TmLRBT) compared with conventional TURBT.

The TmLRBT is increasingly used in the treatment of NMIBC recently, but whether it can provide better cancer control than TURBT is still unclear.

Previous studies have compared the recurrence rates of these two therapies but no significant difference was detected.However, in all these studies, intravesical therapies were conducted using epirubicin or mitomycin C, instead of bacillus Calmette-Guérin (BCG), which is superior for preventing the recurrence of NMIBC.

En-bloc resection of bladder tumor (ERBT) was first described by Kawada et al. in 1997 and has been used by urologists since then. The main advantage of ERBT is that it can resect and extract the entire tumor with a high-quality specimen rather than piecemeal, overcoming some of the short comings of TURBT.

ERBT provides up to 95% of the detrusor muscle, thus leading to a more accurate pathological diagnosis. En-bloc resection is another well recognized procedure that can be performed with various types of energy, such as 2-μm continue-wave laser, holmium laser, Thulium laser, green-light laser, Hybrid-Knife, etc.

The aim of this study is to evaluate and compare the outcome of Thulium laser with the Electrical Trans-urethral en-bloc resection of non-muscle invasive bladder carcinoma regarding efficacy and complications.

ELIGIBILITY:
Inclusion Criteria:

* Age : adults and older adults
* patients with bladder transitional cell carcinoma
* Imaging examinations showed small bladder mass < 3 cm and the bladder muscle has not been affected, no lymph node metastasis or distant metastasis;
* Primary tumor

Exclusion Criteria:

* Large bladder mass > 3 cm measured by CT urography
* Recurrent tumor
* Patients that confirmed post operative histopathology with muscle-invasive bladder transitional cell carcinoma
* Received previous chemotherapy or radiotherapy
* Other pathological types of bladder cancer

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2023-08-13 (Actual); Primary Completion 2024-11-15 (Actual); Study Completion 2024-12-10 (Actual)

PRIMARY OUTCOMES:
Recurrence free survival rate | 12 months
  Number of participants with recurrence free survival during scheduled follow up protocol according to European association of urology guidelines
Local recurrence rate | 12 months
  Number of participants with absence of local recurrence on the site of resection during follow up cystoscopy protocol

SECONDARY OUTCOMES:
Peri-operative complications | Intra operative to 1 week post operative duration
  Number of participants developed peri operative complications regarding severity of bleeding ,number of paricipants developed bladder wall perforation , number of participants developed obturator jerk and severity of lower urinary tract symptoms

CONTACTS AND LOCATIONS:
Overall Officials: Tarek AM Salem, MD, Study Chair — Tarek Abdel magied Salem
Locations (1):
- Helwan university, Helwan, Cairo Governorate, Egypt

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Badawy A, Sultan SM, Marzouk A, El-Sherif E. Thulium laser en bloc resection versus conventional transurethral resection of urinary bladder tumor: A comparative prospective study. Urol Ann. 2023 Jan-Mar;15(1):88-94. doi: 10.4103/ua.ua_59_22. Epub 2022 Nov 8. PMID 37006212